CLINICAL TRIAL: NCT06052384
Title: Optimisation du Parcours de Soins Des Patients Atteints de Douleurs Chroniques : étude randomisée évaluant l'intérêt de l'intégration Des spécialistes du Sommeil
Brief Title: Optimization of the Care Pathway for Patients With Chronic Pain: Assessing the Value of Integrating Sleep Specialists
Acronym: DOLOREPIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RIPH2_PEREZ_DOLOREPIT; 2022-A00919-34 (Other: ID RCB)
Record Dates: First submitted 2023-09-11; First posted 2023-09-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reinforced sleep program (Experimental): standard pain management + sleep disorders management
  Interventions: Other: Standard pain management combined with sleep disorder management
- Standard care (No Intervention): Control group: standard pain management

INTERVENTIONS:
Other: Standard pain management combined with sleep disorder management — Standard pain management combined with sleep disorder management at M6, and M12
  Arms: Reinforced sleep program

SUMMARY:
DOLOREPIT is an interventional, RIPH 2, multicenter, randomized, controlled, open-label study comparing two care pathways for the management of patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* First consultation at the pain management center
* Patient with chronic pain as defined by the "Haute Autorité de Santé". The pain must have several of the following characteristics:

  * Persistence or recurrence
  * Duration beyond what is usual for the presumed initial cause, especially if the pain has been evolving for more than 3 months;
  * Inadequate response to treatment;
  * Important and progressive deterioration of the patient's functional and interpersonal abilities in activities of daily living at home, school, or work due to the pain.
* Patients with chronic primary pain (according to the typology defined by the International Classification of Diseases-11) and classified into one of the 4 following categories:

  * Chronic generalized pain
  * Complex regional pain syndrome
  * Chronic primary headache or orofacial pain
  * Chronic primary musculoskeletal pain
* Pittsburgh Sleep Quality Index (PSQI) must be completed by the patient and the score must be available (for randomization purposes)
* Have access to an internet connection as a self-administered questionnaire is to complete online, and at least have access to the online platform for CBT treatment if insomnia is detected
* Affiliation to a French social security system
* Free informed consent

Exclusion Criteria:

* Patients undergoing cancer treatment or who have completed treatment within the last 2 years
* Patient with a chronic inflammatory disease (e.g. rheumatoid arthritis, ankylosing spondylitis, chronic inflammatory bowel disease, Horton's disease, Wegener's disease, myositis, Still's disease, lupus erythematosus, etc.)
* Immunocompromised patient
* Patient with severe psychiatric pathology that does not allow study follow-up (at the discretion of the investigator)
* Patient already treated for a sleep disorder by a sleep specialist (the only prescription of hypnotics is not considered as a criterion of non-inclusion)
* Patient follow-up difficult (for geographic motives or other reasons)
* Patient under judicial protection of incapable adults or guardianship
* Refusal to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the Mental Composite Score (MCS) of the Short Form 36 Health Survey (SF-36) questionnaire | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  It's a scientifically validated multidimensional scale that provides a generic score for assessing quality of life, regardless of pathology, age or gender. The 36 items of this questionnaire evaluate 8 dimensions: physical activity; limitations due to physical condition; physical pain; perceived health; vitality; life and relationships with others; limitations due to physical condition; psychological health, as well as a separate dimension on the evaluation of perceived health compared to one year earlier. An average score range from 0 to 100 and can be calculated according to an established algorithm. A high score means good health and absence of pain.

SECONDARY OUTCOMES:
The Physical Composite Score (PCS) of the Short Form 36 Health Survey (SF-36) questionnaire | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  It's a scientifically validated multidimensional scale that provides a generic score for assessing quality of life, regardless of pathology, age or gender. The 36 items of this questionnaire evaluate 8 dimensions: physical activity; limitations due to physical condition; physical pain; perceived health; vitality; life and relationships with others; limitations due to physical condition; psychological health, as well as a separate dimension on the evaluation of perceived health compared to one year earlier. An average score range from 0 to 100 and can be calculated according to an established algorithm. A high score means good health and absence of pain.
The score of the French version of the Brief Pain Inventory (BPI). | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  This questionnaire assesses the patient's pain experience and the impact of pain on the patient's daily behavior. It evaluates seven general aspects of the patient's life, divided into fifteen items: activity, mood, walking ability, work, relationships, sleep and enjoyment of life. The score ranges from 0 to 10 with 0 = no pain and 10= worst pain.
The score of the French version of the McGill pain questionnaire (MPQ) | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  This questionnaire assesses the sensory and emotional dimensions of the patient's pain. It is composed of twenty-two items.
  Each item is scored from 0 to 10, with 0 corresponding to "no pain", 5 to "moderate pain" and 10 to "extremely severe pain".
The score of Hospital anxiety and depression scale (HADS) | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  This questionnaire can be used to detect anxiety or depression. For each component (seven items for the "anxiety" component and seven items for the "depression" component), the score obtained is analyzed. A score less than or equal to 7 indicates no symptomatology, a score between 8 and 10 indicates doubtful symptomatology, and a score greater than or equal to 11 indicates definite symptomatology.
The score of the French version of Pittsburgh Sleep Quality Index (PSQI) | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  This is a generic nineteen-item questionnaire for measuring sleep problems. A PSQI score less than or equal to 5 designates "good sleepers", while a score strictly greater than 5 designates "poor sleepers".
The score of the Epworth Sleepiness scale | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  This scale is made up of 8 questions and the final score obtained ranges from 0 to 24: [0-6] = Absence of drowsiness; [7-9] = contentious score which may indicate a pathological condition; [10-24] = Risk of pathological drowsiness.
The score of the Patient Global Impression of Change (PGIC) scale | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  This scale is used to assess the evolution of the patient's state of health in terms of activity limitation, symptoms, emotions and quality of life. This scale ranges from 1 "greatly improved" to 7 "greatly worsened", for which the patient is asked to choose the phrase that best represents the changes in his or her overall health.
The drug consumption, particularly analgesics, antidepressants, benzodiazepines and related hypnotics | Change from baseline (Day 0) at Month 6 (and at Month 12 only for the experimental group)
  INN , dosage and duration
The cost-utility ratio for the medico-economic impact of the care pathway | Change from baseline (Day 0) at Month 6
  The costs avoided in terms of drug consumption, as well as changes in patients' quality of life at different stages.
The score of the International Restless legs syndrome (IRLS) questionnaire | At the 1st sleep consultation (Month 1) then at Month 6 and Month 12
  The latter assesses the severity of RLS according to four levels: for a score between 0 and 10, the disorder is mild; between 11 and 20, moderate; between 21 and 30, severe; between 31 and 40, very severe.
For the experimental group, the average apnea-hypopnea index (AHI) | at start of ventilation (continuous positive airway pressure), then for periods Month 3-Month 6 and Month 6-Month 12
  It represents the average frequency of apneas and hypopneas per hour of sleep. There are three levels of apnea and hypopnea severity. The mild degree corresponds to respiratory incidents of between 5 and 15 per hour, the moderate degree corresponds to respiratory incidents between 15 and 30 per hour, and the severe degree indicates more than 30 respiratory events per hour.
For the experimental group, the score of the insomnia severity index (ISI) | At the 1st sleep consultation (Month 1) then at Month 6 and Month 12
  This validated self-questionnaire consists of 7 questions designed to assess the nature of insomnia, sleep satisfaction, day-to-day functioning and anxiety about sleep disorders. Each of the 7 items is evaluated on a 5-point Likert scale (from 0 to 4). The total score is obtained by adding together the scores of the 7 items . The total score ranges from 0 to 28: [0-7] = No insomnia; [8- 14] = Subclinical insomnia (mild); [15-21] = Clinical insomnia (moderate); [22-28] = Clinical insomnia (severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Emile Roux, Le Puy-en-Velay, France